CLINICAL TRIAL: NCT03756792
Title: Assessing Patient Anxiety During Mohs Micrographic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00054156
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Anxiety
Keywords: Mohs Micographic Surgery; skin cancer; melanoma
MeSH Terms: conditions — Anxiety Disorders; Skin Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First Time Control (Active Comparator): Patients with no prior experience of Mohs surgery will be randomly assigned to the control group. The control group will receive the normal education material that MMS patients receive from Wake Forest Baptist Health Dermatology, then fill out a brief survey.
  Interventions: Behavioral: Normal Education Material
- First Time Intervention (Experimental): Patients with no prior experience of Mohs surgery will be randomly assigned to the intervention group. The intervention group will receive the normal education material that MMS patients receive from Wake Forest Baptist Health Dermatology and read a vignette about the typical experience of a Mohs patient, then fill out a brief survey.
  Interventions: Behavioral: Normal Education Material; Behavioral: Vignette
- Previous Experience Control (Active Comparator): Patients with prior experience of Mohs surgery will be randomly assigned to the control group. The control group will receive the normal education material that MMS patients receive from Wake Forest Baptist Health Dermatology, then fill out a brief survey.
  Interventions: Behavioral: Normal Education Material
- Previous Experience Intervention (Experimental): Patients with prior experience of Mohs surgery will be randomly assigned to the intervention group. The intervention group will receive the normal education material that MMS patients receive from Wake Forest Baptist Health Dermatology and read a vignette about the typical experience of a Mohs patient, then fill out a brief survey.
  Interventions: Behavioral: Normal Education Material; Behavioral: Vignette

INTERVENTIONS:
Behavioral: Normal Education Material — Patients will receive standard educational material about Mohs micrographic surgery.
Behavioral: Vignette — Patients will receive standard educational material about Mohs micrographic surgery and read a vignette detailing the typical experience of a Mohs patient.
  Arms: First Time Intervention; Previous Experience Intervention

SUMMARY:
This study will assess the anxiety that patients are experiencing during a Mohs micrographic surgery. The study will compare the feelings of anxiety experienced by patients returning for Mohs surgery after already undergoing the surgery at least one time to feelings experienced by patients who have never had Mohs surgery before. The study will also compare the feelings experienced by patients who have read a vignette about the typical Mohs experience to the feelings of patients who have not read a vignette.

DETAILED DESCRIPTION:
There has been a continual increase in cases of nonmelanoma skin cancer and melanoma over the last several decades. With the increase in incidence, there is also the need for increased treatment. Mohs micrographic surgery (MMS) is highly efficacious, with cure rates in the upper 90% for both basal cell carcinoma and squamous cell carcinoma, the two most common forms of skin cancer. MMS is used for tumors in cosmetically sensitive areas or areas of recurrence.

While MMS is usually performed in the outpatient setting, it may be an anxiety provoking experience for patients, ranging from the fear of a cancer diagnosis, to concerns about the procedural events of the surgery and associated pain, to the anticipation of their final cosmetic result. During a MMS procedure, unlike many other types of surgery or procedures, the patient is awake and aware of his or her surroundings, with periods of waiting interspersed throughout the procedure. Such aspects can lead to the high level of perioperative anxiety in MMS patients. The effects of listening to music, watching preoperative informational videos, and the use of web-based applications have been used to attempt to decrease anxiety in MMS patients. However, causes for differences in anxiety level between first time MMS patients and patients returning for a subsequent MMS procedure are not well characterized.

One approach to reduce patient anxiety involves patient education, where patients are presented statistics about the small likelihood of complication from the MMS procedure. However, patients interpret these data very subjectively. The study team proposes an alternative approach to patient education through patient vignettes. A previous study explored using a narrative video that included patient testimonials, but this video also used patient-physician interaction and drawings. In this study, patients will be provided short vignettes, that would include information about the experience of a typical MMS patient.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing Mohs micrographic surgery for cutaneous cancer, soft tissue tumors, and adnexal tumors
* Subjects with a working knowledge of English
* Age 18-80

Exclusion Criteria:

* Patients unable to fill out a paper or electronic survey or read a short pamphlet on prior patient experiences, or those unwilling to have either of the previously stated items read aloud to them.
* Individuals less than 18 or greater than 80 years old (line of questioning necessary for the study may be beyond understanding in this group)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Anxiety Scores | up to 10 minutes
  This outcome will assess the difference in VAS-A scores for patients based on prior experience with MMS versus first-time MMS. A higher score denotes a worse outcome.
Visual Analog Scale Scores | up to 10 minutes
  This outcome will assess the difference the difference in VAS-A score between the control and intervention groups that read patient vignettes. A higher score denotes a worse outcome.
Survey to identify factors that modify anxiety - Positive statements | up to 10 minutes
  The survey presents 2 statements to be answered each on a 5-point likert scale to assess patients feelings of anxiety in the perioperative period. A higher score denotes a better outcome. Total score 0-10
Survey to identify factors that modify anxiety - Negative statements | up to 10 minutes
  The survey presents 2 statements to be answered each on a 5-point likert scale to assess patients feelings of anxiety in the perioperative period. A higher score denotes a worse outcome. Total score 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feldman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers HW, Weinstock MA, Feldman SR, Coldiron BM. Incidence Estimate of Nonmelanoma Skin Cancer (Keratinocyte Carcinomas) in the U.S. Population, 2012. JAMA Dermatol. 2015 Oct;151(10):1081-6. doi: 10.1001/jamadermatol.2015.1187. PMID 25928283
- [Background] Dubas LE, Ingraffea A. Nonmelanoma skin cancer. Facial Plast Surg Clin North Am. 2013 Feb;21(1):43-53. doi: 10.1016/j.fsc.2012.10.003. PMID 23369588
- [Background] Kamangar F, Petukhova TA, Monico G, Mathis S, Joo J, Zhuang A, Li CS, Liu Y, Lee E, Eisen D. Anxiety levels of patients undergoing common dermatologic procedures versus those seeking general dermatologic care. Dermatol Online J. 2017 May 15;23(5):13030/qt64d8r1gq. PMID 28537871
- [Background] Persichetti GB, Walling HW, Ceilley RI. Personalized music enhances patient perception of the Mohs surgery experience. Dermatol Surg. 2009 Feb;35(2):265-7. doi: 10.1111/j.1524-4725.2008.34422.x. No abstract available. PMID 19215268
- [Background] Vachiramon V, Sobanko JF, Rattanaumpawan P, Miller CJ. Music reduces patient anxiety during Mohs surgery: an open-label randomized controlled trial. Dermatol Surg. 2013 Feb;39(2):298-305. doi: 10.1111/dsu.12047. Epub 2013 Jan 24. PMID 23346989
- [Background] Newsom E, Lee E, Rossi A, Dusza S, Nehal K. Modernizing the Mohs Surgery Consultation: Instituting a Video Module for Improved Patient Education and Satisfaction. Dermatol Surg. 2018 Jun;44(6):778-784. doi: 10.1097/DSS.0000000000001473. PMID 29642110
- [Background] Hawkins SD, Koch SB, Williford PM, Feldman SR, Pearce DJ. Web App- and Text Message-Based Patient Education in Mohs Micrographic Surgery-A Randomized Controlled Trial. Dermatol Surg. 2018 Jul;44(7):924-932. doi: 10.1097/DSS.0000000000001489. PMID 29406486
- [Background] Zhang J, Miller CJ, O'Malley V, Etzkorn JR, Shin TM, Sobanko JF. Patient quality of life fluctuates before and after Mohs micrographic surgery: A longitudinal assessment of the patient experience. J Am Acad Dermatol. 2018 Jun;78(6):1060-1067. doi: 10.1016/j.jaad.2018.02.065. Epub 2018 Mar 5. PMID 29518455
- [Background] Locke MC, Wilkerson EC, Mistur RL, Nisar M, Love WE. 2015 Arte Poster Competition First Place Winner: Assessing the Correlation Between Patient Anxiety and Satisfaction for Mohs Surgery. J Drugs Dermatol. 2015 Sep;14(9):1070-2. PMID 26355630

DOCUMENTS (1):
  • Informed Consent Form (2020-11-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03756792/ICF_000.pdf